CLINICAL TRIAL: NCT06469242
Title: Clinical Performance of Two Frequent Replacement Silicone Hydrogel Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLM234-C001
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Presbyopia
Keywords: Multifocal; Myopia; Hyperopia
MeSH Terms: conditions — Presbyopia; Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID233309, then Oasys MF (Other): Serafilcon A multifocal contact lenses worn in Period 1, followed by senofilcon A multifocal contact lenses worn in Period 2, as randomized. The study lenses will be worn in a daily wear mode in both eyes (bilaterally) during waking hours for at least 10 hours per day. Each wear period is 14 days (-0/+2). CLEAR CARE will be used for daily cleaning and disinfection.
  Interventions: Device: Serafilcon A multifocal contact lenses; Device: Senofilcon A multifocal contact lenses; Device: CLEAR CARE® Cleaning & Disinfecting Solution
- Oasys MF, then LID233309 (Other): Senofilcon A multifocal contact lenses worn in Period 1, followed by serafilcon A multifocal contact lenses worn in Period 2, as randomized. The study lenses will be worn in a daily wear mode in both eyes (bilaterally) during waking hours for at least 10 hours per day. Each wear period is 14 days (-0/+2). CLEAR CARE will be used for daily cleaning and disinfection.
  Interventions: Device: Serafilcon A multifocal contact lenses; Device: Senofilcon A multifocal contact lenses; Device: CLEAR CARE® Cleaning & Disinfecting Solution

INTERVENTIONS:
Device: Serafilcon A multifocal contact lenses — Investigational multifocal soft contact lenses
  Other Names: LID233309
Device: Senofilcon A multifocal contact lenses — Commercially available multifocal soft contact lenses
  Other Names: ACUVUE® OASYS MULTIFOCAL with PUPIL OPTIMIZED DESIGN; Oasys MF
Device: CLEAR CARE® Cleaning & Disinfecting Solution — Hydrogen peroxide-based contact lens cleaning and disinfection system
  Other Names: CLEAR CARE

SUMMARY:
The purpose of this study is to evaluate the on-eye multifocal clinical performance of investigational LID233309 contact lenses and Oasys multifocal (MF) contact lenses in a daily wear dispensing trial.

DETAILED DESCRIPTION:
Subjects will wear two different contact lens study products in a cross-over fashion. Each study product type will be worn for approximately 14 days. A washout period of 2-4 days will occur prior to the first wear period and between the two wear periods. Subjects will be expected to attend 7 office visits. The total duration of study participation is approximately 40 days with approximately 28 days of lens wear.

ELIGIBILITY:
Key Inclusion Criteria:

* Current wearer of biweekly/monthly replacement multifocal soft contact lenses in both eyes for a minimum of 5 days per week and 10 hours per day during the past 6 months.
* Manifest cylinder equal to or less than 0.75 diopter (D) in each eye.
* Able to wear contact lenses within the available power range with a near ADD of +0.75 D to +2.50 D in each eye.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Currently pregnant or lactating.
* History of amblyopia, strabismus, or binocular vision abnormalities.
* Habitual Oasys MF contact lens wearers or daily disposable contact lens wearers.
* Monovision contact lens wearers and wearers of contact lens in one eye only.
* Other protocol-defined exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Kurata Eyecare Center, Los Angeles, California
  - Elsa Pao, OD, Oakland, California
  - Drs. Giedd, P.A., Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Wesley Optometric Consulting, Medina, Minnesota
  - ProCare Vision Centers, Inc., Granville, Ohio
  - Insight Research Clinic LLC, Powell, Ohio
  - Optometry Group, PLLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 8 investigative sites.
Pre-assignment Details: Of the 106 subjects enrolled, 2 subjects were discontinued prior to exposure to the study product. This reporting group population includes all subjects exposed to any study lenses evaluated in this study.
Groups:
- LID233309, Then Oasys MF: Serafilcon A multifocal contact lenses worn in Period 1, followed by senofilcon A multifocal contact lenses worn in Period 2, as randomized. The study lenses were worn in a daily wear mode both eyes (bilaterally) during waking hours for at least 10 hours per day. Each wear period was 14 days (-0/+2). CLEAR CARE was used for daily cleaning and disinfection.
- Oasys MF, Then LID233309: Senofilcon A multifocal contact lenses worn in Period 1, followed by serafilcon A multifocal contact lenses worn in Period 2, as randomized. The study lenses were worn in a daily wear mode in both eyes (bilaterally) during waking hours for at least 10 hours per day. Each wear period was 14 days (-0/+2). CLEAR CARE was used for daily cleaning and disinfection.
Period: First Wear Period (Approx 14 Days)
Arm/Group | LID233309, Then Oasys MF | Oasys MF, Then LID233309
Started | 53 | 51
Completed | 48 | 47
Not Completed | 5 | 4
Not completed — Protocol Violation | 4 | 3
Not completed — As Per Sponsor Guidance | 1 | 1
Period: Second Wear Period (Approx 14 Days)
Arm/Group | LID233309, Then Oasys MF | Oasys MF, Then LID233309
Started | 48 | 47
Completed | 48 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects exposed to any study lenses evaluated in this study.
Groups:
- LID233309, Then Oasys MF: Serafilcon A multifocal contact lenses worn in Period 1, followed by senofilcon A multifocal contact lenses worn in Period 2, as randomized. The study lenses were worn in a daily wear mode in both eyes (bilaterally) during waking hours for at least 10 hours per day. Each wear period was 14 days (-0/+2). CLEAR CARE was used for daily cleaning and disinfection.
- Total: Total of all reporting groups
Arm/Group | LID233309, Then Oasys MF | Oasys MF, Then LID233309 | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (7.0) | 53.5 (6.7) | 52.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 18 | 14 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  White | 37 | 37 | 74
  Black or African American | 2 | 1 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 11 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 1 | 1
  Multi-Racial | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 50 | 49 | 99
Region of Enrollment [Number; unit: participants]
  United States | 53 | 51 | 104

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular Visual Acuity at Distance (4 Meters) at Week 1
Description: Visual Acuity (VA) was assessed at a distance of 4 meters with both eyes together (binocular) under high contrast, high illumination lighting with study lenses in place. VA was measured using letter charts and recorded in the logarithm of the minimum angle of resolution (LogMAR). A LogMAR value of 0 equates to 20/20 Snellen VA (normal distance eyesight), with negative LogMAR values representing better than 20/20 VA. The LogMAR VA scale ranges from -0.30 (20/10 Snellen) to 1.00 (20/200 Snellen). No hypothesis testing was pre-specified for this endpoint.
Time Frame: Week 1 (Day 7 -0/+1 days) of each wear period. A wear period was 14 days (-0/+2 days) according to randomization assignment.
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- LID233309: Serafilcon A multifocal contact lenses worn in Period 1 or Period 2, as randomized. The study lenses were worn in a daily wear mode both eyes (bilaterally) during waking hours for at least 10 hours per day for 14 days (-0/+2). CLEAR CARE was used for daily cleaning and disinfection.
- Oasys MF: Senofilcon A multifocal contact lenses worn in Period 1 or Period 2, as randomized. The study lenses were worn in a daily wear mode in both eyes (bilaterally) during waking hours for at least 10 hours per day for 14 days (-0/+2). CLEAR CARE was used for daily cleaning and disinfection.
Arm/Group | LID233309 | Oasys MF
Number analyzed (Participants) | 99 | 97
logMAR | -0.08 (0.09) | -0.08 (0.09)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, approximately 40 days. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects exposed to any study lenses evaluated in this study, as treated.
Description: All subjects were monitored for serious and other ocular and nonocular AEs. However, the nonocular AE arms were not considered at Risk for ocular adverse event terms as the arms are reporting nonocular-specific AEs. Similarly, the ocular AE arms were not considered at Risk for nonocular adverse event terms as the arms are reporting ocular-specific AEs. All-Cause Mortality was not monitored for the ocular arms.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study lenses.
- LID233309 Ocular; LID233309 Nonocular: Events reported in this group occurred while exposed to the serafilcon A multifocal contact lenses.
- Oasys MF Ocular; Oasys MF Nonocular: Events reported in this group occurred while exposed to the senofilcon A multifocal contact lenses.
Arm/Group | Pretreatment | LID233309 Ocular | LID233309 Nonocular | Oasys MF Ocular | Oasys MF Nonocular
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/0 | 0/100 | 0/0 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/200 | 0/100 | 0/198 | 0/99
Other Adverse Events (participants affected / at risk) | 0/104 | 0/200 | 0/100 | 0/198 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT06469242/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT06469242/SAP_001.pdf